CLINICAL TRIAL: NCT06919094
Title: A Virtual Life Story Club Intervention to Improve Loneliness and Apathy in Community-Dwelling Older Adults: A Mixed-Methods Feasibility Study
Brief Title: A Virtual Life Story Club Intervention to Improve Loneliness and Apathy in Community-Dwelling Older Adults
Acronym: LSC Feasible
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-16787; UM1TR004400 (NIH)
Record Dates: First submitted 2025-03-26; First posted 2025-04-09 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Apathy; Loneliness; Reminiscence Therapy
Keywords: Apathy; Social Isolation; Loneliness; Reminiscence Therapy
MeSH Terms: conditions — Lethargy; Social Isolation

STUDY DESIGN:
Intervention Model Description: Reminiscence therapy will be provided by the Life Story Club©. Participants will meet virtually via Zoom© with their group (6-10 people) weekly for one hour over a 12-week period to exchange life stories and share in conversation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Life Story Club (Experimental): Virtual Group Reminiscence Therapy
  Interventions: Behavioral: Life Story Club

INTERVENTIONS:
Behavioral: Life Story Club — Virtual group reminiscence therapy will be provided by the Life Story Club©. Participants will meet virtually via Zoom© with their group (6-10 people) weekly for one hour over a 12-week period to exchange life stories and share in conversation. Groups will be conducted in entirely in English or Spanish, based on participant preference. Each week, the LSC© facilitator will guide the group with question prompts to encourage participants to share personal information, build friendships & rapport, and create a sense of community. LSC© facilitators are trained in group interview techniques, technology management, and know how to respond appropriately to sensitive information that may emerge during group exchanges.

SUMMARY:
Reminiscence therapy is a non-invasive, non-pharmacological intervention that has been shown to improve cognition, mood, functional status, quality of life, and apathy in older adults. Group reminiscence therapy combines structured social engagement and recounting of personal stories that address both social connection (a risk factor for cognitive decline) and cognition. Life story club© (LSC) is an established, non-profit organization that provides virtual, group reminiscence therapy for older adults to reduce loneliness and promote a sense of belonging and has not been formally studied.

DETAILED DESCRIPTION:
The purpose of this study is to explore the feasibility of a LSC© intervention to improve loneliness and apathy in community-dwelling older adults.

This pilot study will be conducted to compare loneliness and apathy in lonely individuals without dementia at baseline who receive a virtual group reminiscence therapy intervention (vGRT). The intervention will be delivered weekly over 12 weeks. Loneliness and apathy will be assessed before and after the intervention as described in the Outcome Measures section of this registration. Feasibility will be assessed using quantitative and qualitative measures including feasibility of screening and enrollment, acceptability, and program satisfaction. Qualitative interviews will be conducted with a subset of 30 individuals to explore acceptability, barriers, and facilitators of the intervention.

This study will provide evidence for the feasibility of a virtual group reminiscence therapy for community dwelling older adults to reduce loneliness and apathy. This approach is both innovative and pragmatic because it will leverage an existing community-based service, with an established infrastructure and track record within the community to deliver the intervention. As such, the proposed research has the potential for broad implications for community-based research and aligns with multiple translational science principles.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 and over
* English or Spanish fluency
* Able to provide informed consent

Exclusion Criteria:

* Dementia based on Aging and Dementia (AD8) score of ≥4 or previous dementia diagnosis
* Severe auditory or visual loss
* Lack of access to internet connection or phone

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Loneliness | From baseline to 3 months and 6 months
  Loneliness will be assessed using the University of California, Los Angeles (UCLA) Loneliness Scale questionnaire. The UCLA Loneliness Scale is a 20-item measure that assesses how often a person feels disconnected from others. Participants provide responses using a 4-point Likert scale where 1 = never; 2 = rarely; 3 = sometimes; 4 = always, for an overall possible scoring range of 20-80, such that higher scores are associated with increased loneliness. Positively worded items in the questionnaire must be reverse-coded before reporting. For purposes of this study changes from baseline to 3 months and baseline to 6 months will be assessed whereby positive values are indicative of an increase in loneliness from baseline and negative values a decrease in loneliness from baseline. Group scores will be summarized using basic descriptive statistics.
Change in Apathy | From baseline to 3 months and 6 months
  Apathy will be assessed using the self-reported Apathy Evaluation Scale (AES-S). The AES-S is an 18-item questionnaire that addresses characteristics of goal directed behavior that reflects apathy including behavioral, cognitive, and emotional indicators. Participants provide responses based on a 4-point Likert scale where 1 = not at all true; 2 = slightly true; 3 = somewhat true; and 4 = very true, for an overall possible scoring range of 18-72, such that higher scores are associated with greater apathy. Positively worded items in the scale must be reverse-coded before reporting. For purposes of this study changes from baseline to 3 months and baseline to 6 months will be assessed whereby positive values are indicative of increased apathy from baseline and negative values decreased apathy from baseline. Group scores will be summarized using basic descriptive statistics.

SECONDARY OUTCOMES:
Change in cognition | From baseline to 3 months and 6 months
  Cognition will be assessed using a version of the Telephone-Montreal Cognitive Assessment (T-MoCA). The T-MoCA is a 22-item phone-administered exam which assesses a range of global cognitive domains including attention, memory, language, and orientation. Each item is one point yielding an overall possible scoring range of 0-22, with higher scores being indicative of better cognitive function. Scores of 18 or below are generally suggestive of Mild Cognitive Impairment (MCI). For purposes of this study changes from baseline to 3 months and baseline to 6 months will be assessed whereby positive values are indicative of increased cognition from baseline and negative values decreased cognition from baseline. Group scores will be summarized using basic descriptive statistics. To reduce practice effect Version (V)8.1 will be administered at baseline, V8.2 at 3 months, and V8.3 at 6 months. Scoring ranges are identical for all 3 versions.
Change in Depressive Symptoms | From baseline to 3 months and 6 months
  Depressive symptoms will be assessed by administration of the Geriatric Depression Scale - Short Form (GDS-15), The GDS-15 is a 15-item questionnaire in which participants provide a dichotomous (Yes/No) response as to how they have felt over the prior week. Answers suggestive of depression are bolded/italicized on the questionnaire (may either be 'Yes' or 'No' depending on the item). A score of 1 point is assigned for each bolded/italicized response such that higher scores are associated with more depressive symptoms. A score of 0 to 5 is normal. A score greater than 5 suggests depression. For purposes of this study changes from baseline to 3 months and baseline to 6 months will be assessed whereby positive values are indicative of increase in depressive symptoms from baseline and negative values a decrease in depressive symptoms from baseline. Results will be summarized using basic descriptive statistics.
Change in Meaning and Purpose | From baseline to 3 months and 6 months
  Meaning and purpose will be assessed as a composite measure using the Patient-Reported Outcomes Measurement Information System (PROMIS) Meaning and Purpose 4-item scale. The 4-item scale is designed to assess an individual's subjective experience of meaning and purpose in life. Participants provide responses on a 5-point Likert scale ranging from 1-5 for an overall possible scoring range of 4-20, such that higher scores are associated with greater meaning and purpose. For purposes of this study changes from baseline to 3 months and baseline to 6 months will be assessed whereby positive values are indicative of increased experiences of meaning and purpose from baseline and negative values decreased experiences of meaning and purpose from baseline. Group results will be summarized using basic descriptive statistics
Change in Social Support | From baseline to 3 months and 6 months
  Social Support will be assessed using the Medical Outcomes Study (MOS) Social Support Scale. The MOS is a 19-item multidimensional, self-administered instrument that measures the availability of support, if needed. The overall social support component of the MOS Social Support scale will be used. Participants provide responses on a 5-point Likert scale ranging from 1-5 for an overall possible scoring range of 19-95, such that higher scores are associated with greater availability of social support. For purposes of this study changes from baseline to 3 months and baseline to 6 months will be assessed whereby positive values are indicative of increased social support and purpose from baseline and negative values decreased social support from baseline. Group results will be summarized using basic descriptive statistics

CONTACTS AND LOCATIONS:
Overall Officials: Mirnova Ceide, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing to be determined.

REFERENCES:
- [Background] Allen AP, Doyle C, Roche RAP. The Impact of Reminiscence on Autobiographical Memory, Cognition and Psychological Well-Being in Healthy Older Adults. Eur J Psychol. 2020 May 29;16(2):317-330. doi: 10.5964/ejop.v16i2.2097. eCollection 2020 May. PMID 33680185
- [Background] Choy JCP, Lou VWQ. Effectiveness of the Modified Instrumental Reminiscence Intervention on Psychological Well-Being Among Community-Dwelling Chinese Older Adults: A Randomized Controlled Trial. Am J Geriatr Psychiatry. 2016 Jan;24(1):60-69. doi: 10.1016/j.jagp.2015.05.008. Epub 2015 May 19. PMID 26419735
- [Background] Cuevas PEG, Davidson PM, Mejilla JL, Rodney TW. Reminiscence therapy for older adults with Alzheimer's disease: A literature review. Int J Ment Health Nurs. 2020 Jun;29(3):364-371. doi: 10.1111/inm.12692. Epub 2020 Jan 26. PMID 31984570
- [Background] Kirk M, Rasmussen KW, Overgaard SB, Berntsen D. Five weeks of immersive reminiscence therapy improves autobiographical memory in Alzheimer's disease. Memory. 2019 Apr;27(4):441-454. doi: 10.1080/09658211.2018.1515960. Epub 2018 Sep 8. PMID 30198380
- [Background] Platel H, Eustache ML, Coppalle R, Viard A, Eustache F, Groussard M, Desgranges B. Boosting Autobiographical Memory and the Sense of Identity of Alzheimer Patients Through Repeated Reminiscence Workshops? Front Psychol. 2021 Feb 15;12:636028. doi: 10.3389/fpsyg.2021.636028. eCollection 2021. PMID 33679562
- [Background] Syed Elias SM, Neville C, Scott T. The effectiveness of group reminiscence therapy for loneliness, anxiety and depression in older adults in long-term care: a systematic review. Geriatr Nurs. 2015 Sep-Oct;36(5):372-80. doi: 10.1016/j.gerinurse.2015.05.004. Epub 2015 Jun 19. PMID 26099638
- [Background] Saragih ID, Tonapa SI, Yao CT, Saragih IS, Lee BO. Effects of reminiscence therapy in people with dementia: A systematic review and meta-analysis. J Psychiatr Ment Health Nurs. 2022 Dec;29(6):883-903. doi: 10.1111/jpm.12830. Epub 2022 Apr 17. PMID 35348260
- [Background] Lok N, Bademli K, Selcuk-Tosun A. The effect of reminiscence therapy on cognitive functions, depression, and quality of life in Alzheimer patients: Randomized controlled trial. Int J Geriatr Psychiatry. 2019 Jan;34(1):47-53. doi: 10.1002/gps.4980. Epub 2018 Sep 24. PMID 30246408